CLINICAL TRIAL: NCT03930394
Title: Vascular Cardiotoxicity of Ponatinib
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Assistant Professor, Oregon Health and Science University
Other Study IDs: Ponatinib Cardiotoxicity
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Cardiotoxicity
MeSH Terms: conditions — Cardiotoxicity | interventions — Ultrasonography, Carotid Arteries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Contrast ultrasound perfusion imaging — Contrast ultrasound perfusion imaging for microvascular perfusion, and carotid ultrasound data on intima-media thickness (or plaque size) will be serially assessed in subjects started on ponatinib.
  Other Names: Carotid ultrasound

SUMMARY:
Pre-clinical studies suggest that the third generation tyrosine kinase inhibitor ponatinib can result in microvascular angiopathy and acceleration of atherosclerosis. This study is intended to examine for myocardial microvascular angiopathy and changes in carotid plaque in patients receiving ponatinib as part of their clinical care.

DETAILED DESCRIPTION:
In this study, we will perform serial echocardiography for ventricular function, myocardial contrast echocardiography for microvascular perfusion assessment, blood analysis for myocardial injury, and carotid US for plaque or IMT progression in subjects receiving ponatinib. This series of tests is intended to provide information on the presence of clinically-evident or subclinical microvascular angiopathy and plaque acceleration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CML or ALL
* Prescribed ponatinib

Exclusion Criteria:

* pregnancy or lactation
* major medical illness involving the heart or vasculature (CAD, PAD, DCM).
* hemodynamically unstable
* allergy to ultrasound contrast agents.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with CML or ALL who are to be treated with ponatinib.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Presence versus absence of any myocardial perfusion defect assessed by visual analysis for any abnormalities of microvascular flux rate (beta function) or microvascular blood volume during an infusion of ultrasound microbubble contrast agents. | 6 months
  Contrast ultrasound perfusion imaging will be performed using power-modulation imaging and infusion of an ultrasound contrast agent. Destruction replenishment kinetics will be assessed visually by examination of delayed replenishment of signal intensity (>5 seconds) after a high-mechanical index burst sequence, or abnormalities in plateau intensity reflecting regional abnormalities in myocardial microvascular blood volume.
Presence versus absence of any myocardial perfusion defect assessed by visual analysis for any abnormalities of microvascular flux rate (beta function) or microvascular blood volume during an infusion of ultrasound microbubble contrast agents. | 12 months
  Contrast ultrasound perfusion imaging will be performed using power-modulation imaging and infusion of an ultrasound contrast agent. Destruction replenishment kinetics will be assessed visually by examination of delayed replenishment of signal intensity (>5 seconds) after a high-mechanical index burst sequence, or abnormalities in plateau intensity reflecting regional abnormalities in myocardial microvascular blood volume.
Carotid plaque size | 6 months
  Changes in IMT or plaque size
Carotid plaque size | 12 months
  Changes in IMT or plaque size

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon HSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Latifi Y, Moccetti F, Wu M, Xie A, Packwood W, Qi Y, Ozawa K, Shentu W, Brown E, Shirai T, McCarty OJ, Ruggeri Z, Moslehi J, Chen J, Druker BJ, Lopez JA, Lindner JR. Thrombotic microangiopathy as a cause of cardiovascular toxicity from the BCR-ABL1 tyrosine kinase inhibitor ponatinib. Blood. 2019 Apr 4;133(14):1597-1606. doi: 10.1182/blood-2018-10-881557. Epub 2019 Jan 28. PMID 30692122